CLINICAL TRIAL: NCT01305694
Title: PhaseⅠ/ⅡTrial of Bone Marrow Derived Mesenchymal Stem Cell Transplantation From Related Donor to Patients With Relapsed/Refractory Aplastic Anemia.
Brief Title: Mesenchymal Stem Cells Transplantation to Patients With Relapsed/Refractory Aplastic Anemia.
Acronym: MSC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Guangzhou Municipal Twelfth People's Hospital (Other); Guangdong Prevention and Treatment Center for Occupational Diseases (Other)
Responsible Party: Jian Liu (President of the hospital), Guangzhou General Hospital of Guangzhou Military Command
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-2010-16
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2011-02

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MSC (Experimental): Intravenous bone marrow derived mesenchymal stem cells infusion from related donor to patients with relapsed/refractory aplastic anemia.
  Interventions: Biological: bone marrow derived mesenchymal stem cells

INTERVENTIONS:
Biological: bone marrow derived mesenchymal stem cells — Intravenous administration of up to 6x10^5 MSCs per kg,qw,for 4 weeks
  Other Names: Mesenchymal Stem Cells; Multipotent Mesenchymal Stem Cells; Multipotent Mesenchymal Stromal Cells

SUMMARY:
The study is a phase I/II trial designed to establish the safety and efficacy of intravenous administration of bone marrow derived mesenchymal stem cells from related donor to patients with relapsed/refractory aplastic anemia.

DETAILED DESCRIPTION:
Aplastic anemia (AA) is an autoimmune hematologic stem cell disease mediated by activated T-lymphocytes that leads to bone marrow dysfunction. In the presence of an empty marrow, pancytopenia, and transfusion dependence, the severity of the disease is based on neutrophil (PMN) count: nonsevere AA (nSAA; PMN > 0.5 × 109/L), severe AA (SAA;PMN 0.2- 0.5 × 109/L), and very severe AA (vSAA; PMN< 0.2 × 109/L). Patients with nSAA can be offered supportive care, anabolic steroids, and/or low-dose steroids or cyclosporine (CsA).Patients with SAA and vSAA can be offered immunosuppressive treatment involving injections of Anti-thymocyte globulin (ATG) in combination with cyclosporine (CsA). However, some nSAA patients remains dependent to transfusion, the treatment response with ATG for SAA is at best between 50-60%,30%-40% patients relapse following an initial response to treatment, they also do not have a HLA-matched donor for bone marrow transplantation. These patients have a high risk of dying without additional treatment. Since the prognosis of these refractory and relapsed AA patients remains poor, there is a need for more safe and effective therapy that can improve response rates and remission duration in refractory and relapsed AA.

Mesenchymal stem cells (MSCs) are part of the bone marrow stem cells repertoire. The main role of MSCs is to support hematopoiesis. Recently, significant interactions between MSCs and cells from the immune system have been demonstrated:MSCs were found to downregulate T and B lymphocytes, natural killer cells (NK) and antigen presenting cells through various mechanisms, including cell-to-cell interaction and soluble factor production. MSCs can fully suppress T cell function which involves some degree of MSC activation or 'licensing' thought to involve interferon (IFN)-γ in conjunction with IL-1α, IL-1β or tumour necrosis factor-a. Non-specific suppression of T cell proliferation is mediated by soluble factors such as transforming growth factor (TGF)-β, kynurenine, prostaglandin E2 (PGE2), nitric oxide, haem oxygenase products and insulin-like growth factor binding protein. Since the haematopoietic support and immunomodulatory effects, bone marrow-derived human MSCs transplantation maybe a safe novel therapeutic approach for patients with refractory and relapsed AA.

ELIGIBILITY:
Inclusion Criteria:

* Patients must fulfill definition of aplastic anaemia:

There must be at least two of the following:

haemoglobin < 100g/L; platelet count < 50 x 109/L; neutrophil count < 1.5 x 109/L, and a hypocellular bone marrow;

SAA as defined by a hypocellular bone marrow of <25% cellularity and two of the following:

neutrophil count < 0.5 x 109/L platelets < 20 x 109/L reticulocytes < 20 x 109/L nSAA as defined by a hypocellular bone marrow and cytopenia in at least two cell lines and neutrophil count > 0.5 x 109/L, and red cell and/or platelet transfusion dependence.

* Patients belong to acquired aplastic anaemia.
* Patients with a history SAA must have had an incomplete response at least 3 months following treatment with ATG/CsA, or they must have relapsed following an initial response to treatment, and they do not have a HLA-matched donor for bone marrow transplantation. Patients with a history nSAA must have red cell and/or platelet transfusion dependence.
* Peripheral blood counts at the time of enrollment must include at least one of the following: haemoglobin < 90 g/L or red blood cell (RBC) transfusion dependence, PMN < 1 x 109/L, or platelet count < 50 x 109/L.
* Patients must have organ function as defined below:

total bilirubin within normal institutional limits (NV: 0.0-20.5 umol/L) AST(SGOT)/ALT(SGPT) < 2.5 × institutional upper limit of normal AST (NV: 0-35 U/L); ALT (NV: 0-40 U/L) Creatinine within normal institutional limits (NV: 53-106 umol/L) or Creatinine clearance > 1.25 ml/s for patients with creatinine levels above institutional normal.

* Age minimum 16 years old with no upper age limit.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents within 4 weeks of study entry.
* History of allergic reactions attributed to compounds of similar biologic composition to mesenchymal stem cells.
* Current diagnosis of Fanconi's anemia, Dyskeratosis Congenita (DC) or other hereditary forms of AA.
* Psychiatric, addictive or any other disorder that compromises ability to give a truly informed consent.
* Age < 16 years old.
* ECOG performance status > 2.
* Malignancy within the last 5 years.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (defined as invasive fungal infection and progressive CMV viremia), symptomatic congestive heart failure (NYH class III and IV), unstable angina pectoris, or cardiac arrhythmia.
* Pregnant or breastfeeding women.
* HIV-positive patients.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | up to 30 days

SECONDARY OUTCOMES:
Hematologic response | up to 1 year
Relapse | up to 1 year
Clonal evolution to PNH, myelodysplasia or acute leukemia | up to 1 year
Survival | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yang Xiao, MD, Study Director — Guangzhou General Hospital of Guangzhou Military Command
Locations (1):
- Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bacigalupo A. Aplastic anemia: pathogenesis and treatment. Hematology Am Soc Hematol Educ Program. 2007:23-8. doi: 10.1182/asheducation-2007.1.23. PMID 18024605
- [Background] Di Nicola M, Carlo-Stella C, Magni M, Milanesi M, Longoni PD, Matteucci P, Grisanti S, Gianni AM. Human bone marrow stromal cells suppress T-lymphocyte proliferation induced by cellular or nonspecific mitogenic stimuli. Blood. 2002 May 15;99(10):3838-43. doi: 10.1182/blood.v99.10.3838. PMID 11986244
- [Background] Polchert D, Sobinsky J, Douglas G, Kidd M, Moadsiri A, Reina E, Genrich K, Mehrotra S, Setty S, Smith B, Bartholomew A. IFN-gamma activation of mesenchymal stem cells for treatment and prevention of graft versus host disease. Eur J Immunol. 2008 Jun;38(6):1745-55. doi: 10.1002/eji.200738129. PMID 18493986
- [Background] English K, Barry FP, Field-Corbett CP, Mahon BP. IFN-gamma and TNF-alpha differentially regulate immunomodulation by murine mesenchymal stem cells. Immunol Lett. 2007 Jun 15;110(2):91-100. doi: 10.1016/j.imlet.2007.04.001. Epub 2007 Apr 26. PMID 17507101
- [Background] Ryan JM, Barry F, Murphy JM, Mahon BP. Interferon-gamma does not break, but promotes the immunosuppressive capacity of adult human mesenchymal stem cells. Clin Exp Immunol. 2007 Aug;149(2):353-63. doi: 10.1111/j.1365-2249.2007.03422.x. Epub 2007 May 22. PMID 17521318
- [Background] Aggarwal S, Pittenger MF. Human mesenchymal stem cells modulate allogeneic immune cell responses. Blood. 2005 Feb 15;105(4):1815-22. doi: 10.1182/blood-2004-04-1559. Epub 2004 Oct 19. PMID 15494428
- [Background] Sato K, Ozaki K, Oh I, Meguro A, Hatanaka K, Nagai T, Muroi K, Ozawa K. Nitric oxide plays a critical role in suppression of T-cell proliferation by mesenchymal stem cells. Blood. 2007 Jan 1;109(1):228-34. doi: 10.1182/blood-2006-02-002246. Epub 2006 Sep 19. PMID 16985180
- [Background] Chabannes D, Hill M, Merieau E, Rossignol J, Brion R, Soulillou JP, Anegon I, Cuturi MC. A role for heme oxygenase-1 in the immunosuppressive effect of adult rat and human mesenchymal stem cells. Blood. 2007 Nov 15;110(10):3691-4. doi: 10.1182/blood-2007-02-075481. Epub 2007 Aug 7. PMID 17684157
- [Background] Gieseke F, Schutt B, Viebahn S, Koscielniak E, Friedrich W, Handgretinger R, Muller I. Human multipotent mesenchymal stromal cells inhibit proliferation of PBMCs independently of IFNgammaR1 signaling and IDO expression. Blood. 2007 Sep 15;110(6):2197-200. doi: 10.1182/blood-2007-04-083162. Epub 2007 May 23. PMID 17522338
- [Background] Kassis I, Vaknin-Dembinsky A, Karussis D. Bone marrow mesenchymal stem cells: agents of immunomodulation and neuroprotection. Curr Stem Cell Res Ther. 2011 Mar;6(1):63-8. doi: 10.2174/157488811794480762. PMID 20955154
- [Derived] Xiao Y, Jiang ZJ, Pang Y, Li L, Gao Y, Xiao HW, Li YH, Zhang H, Liu Q. Efficacy and safety of mesenchymal stromal cell treatment from related donors for patients with refractory aplastic anemia. Cytotherapy. 2013 Jul;15(7):760-6. doi: 10.1016/j.jcyt.2013.03.007. PMID 23731760